CLINICAL TRIAL: NCT05080465
Title: Long Term Follow up Autologous Mesenchymal Stem Cell Therapy for Patients Virus-related Liver Cirrhosis
Brief Title: Long Term Follow up Mesenchymal Stem Cell Therapy for Patients Virus-related Liver Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ukraine Association of Biobank (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAB00240818-1
Record Dates: First submitted 2019-08-29; First posted 2021-10-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Fibrosis; Pathologic Processes; Liver Diseases; Digestive System Diseases; Stem Cell; MSC Therapy; Mesenchymal
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Pathologic Processes; Liver Diseases; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: As the primary objective of the study is to assess safety of MSC infusion, a single arm non-blinded study design has been adopted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A single dose of 0.5 to 1 x 10^6/kg autologous BM MSCs (Total volume: 30 - 50 ml) will be infused via peripheral venous access.
  Interventions: Biological: Autologous BM MSC

INTERVENTIONS:
Biological: Autologous BM MSC — A total of 100-200ml will be harvested from the subject, in either a single or multiple punctures. This will be processed for autologous MSC infusion.

SUMMARY:
This is a study to assess safety and preliminary clinical activity of treatments of liver cirrhosis in patients with caused by Hepatitis C and Hepatitis B or Nonalcoholic Steatohepatitis of Mesenchymal stem cell.

Patients who will be enrolled in the study will be under supervision and monitoring to ensure clinical significance

DETAILED DESCRIPTION:
Liver cirrhosis refers to extreme scarring of the liver, resulting in suboptimal function of the liver. It can result from a variety of causes, ranging from hepatitis B and C infection, excessive alcohol consumption, autoimmune causes, fatty liver and others. Irrespective of the cause, once the liver becomes cirrhotic, it is a downhill course.

Liver cirrhosis is irreversible and most patients will progressively worsen over time. Once liver cirrhosis has reached the stage of decompensation, that is, development of jaundice, ascites, variceal bleeding, hepatic encephalopathy and coagulopathy the two-year survival drops to about 50%.

The definitive treatment of decompensated cirrhosis is liver transplantation. While a liver transplantation is potentially curative, the high costs, lack of a donor, treatment-related mortality and the immunosuppression complications make this option possible only for a limited number of patients. The vast majority do not have an effective option at all, thus the need to develop alternative therapies. Various types of Stem Cells had been investigated as a regenerative therapy for liver cirrhosis. These stem cells include bone marrow mesenchymal stem cells (MSC). Some early studies have shown encouraging results in patients who had autologous bone marrow stem cell transplantation. There was improved liver function in these patients with cirrhotic livers.

The sponsor is proposing a study to look into the role of MSC therapy for patients with liver cirrhosis in Ukraine. This will be a Phase I study with the main emphasis on the safety and efficiency profile first. The trial will be conducted in compliance with the protocol, GCP and local regulatory requirement(s).

ELIGIBILITY:
Inclusion Criteria:

Provision of written informed consent for this study by subject or as applicable legal guardians Able to comply with study requirements Еру rates with RVR defined as serum HCV RNA undetectable after 12 month after antiviral therapy.

Subject must have documented compensated cirrhosis and no current or past clinical evidence of decompensated liver disease Subject must have documented history Screening laboratory result indicating hepatitis C virus (HCV) Genotype 1, 2, 4, 5 or 6 (GT1,2,4,5,6) infection

Exclusion Criteria:

Positive test result at screening for Hepatitis B surface antigen or anti-human immunodeficiency virus (anti-HIV) antibody HCV genotype performed during screening indicating co-infection with more than 1 HCV genotype.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
MR Elastography | Change from Baseline (Day 0) until 40 weeks
  The detect liver stiffness of significant or severe fibrosis (≥stage F2)\(≥stage F3)
The level of serum alanine aminotransferase (ALT) | Change from Baseline (Day 0) until 40 weeks
  level of serum alanine aminotransferase less 40 (IU/L)
Clinical Examination | Change from Baseline (Day 0) until 40 weeks
  To observe for the following:
  absence of grade IV anaphylactic reactions (in reference to CTCAE 4.03)
The level of glomerular filtration rate (GFR) | Change from Baseline (Day 0) until 40 weeks
  The level of glomerular filtration range from 90 to 120 mL/min/1.73 m2

SECONDARY OUTCOMES:
The level of serum albumin (ALB) | Up to 6 months, post-infusion
  The level of serum albumin to 5.4 g/dL
The level of serum total bilirubin (TB) | Up to 6 months, post-infusion
  The level of serum total bilirubin 1.8 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Bio-Stem Cell Rehabilitation, Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: No